CLINICAL TRIAL: NCT00612573
Title: Phase 2 Study Randomized, Double-blind Study to Evaluate the Safety and Efficacy of 3 Doses of Doxycycline as Compared to Placebo in the Treatment of Moderate to Severe Facial Acne Vulgaris
Brief Title: Treatment of Moderate to Severe Facial Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-07907; WC2055
Record Dates: First submitted 2008-01-25; First posted 2008-02-11 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Doxycyline 0.6 mg/kg/day (Experimental): Doxycycline dosed at 40 mg/day to subjects of appropriate weights
  Interventions: Drug: Doxycycline 0.6 mg/kg/day
- Doxycycline 1.2 mg/kg/day (Experimental): Doxycycline dosed at 80 mg/day to subjects of appropriate weights
  Interventions: Drug: Doxycycline 1.2 mg/kg/day
- Doxycycline 2.4 mg/kg/day (Experimental): Doxycycline dosed at 160 mg/day to subjects of appropriate weights
  Interventions: Drug: Doxycycline 2.4 mg/kg/day
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline 0.6 mg/kg/day — doxycycline 40 mg/day, oral, 12 weeks
  Arms: Doxycyline 0.6 mg/kg/day
Drug: Doxycycline 1.2 mg/kg/day — doxycycline 80 mg/day, 12 weeks
  Arms: Doxycycline 1.2 mg/kg/day
Drug: Doxycycline 2.4 mg/kg/day — doxycycline 160 mg/day, 12 weeks
  Arms: Doxycycline 2.4 mg/kg/day
Drug: Placebo — Placebo, 12 weeks
  Arms: Placebo

SUMMARY:
Randomized, multi-center, double-blind, placebo-controlled 12-week study to assess the safety and efficacy of 3 doses of an oral formulation of Doxycycline oral tablets using the Investigator's Global Assessment (IGA) score and the absolute change from baseline in inflammatory lesion count in patients with moderate to severe facial acne vulgaris. Additionally, the absolute change from baseline in non-inflammatory and total lesions of the active study medication to placebo will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 12 and 45 years of age.
* Has a diagnosis of moderate to severe facial acne vulgaris with no more than two nodules on the face

Exclusion Criteria:

* Is allergic to tetracycline-class antibiotics or to any ingredient in the study medication.
* Has a history of pseudomembranous colitis or antibiotic-associated colitis.
* Has a history of hepatitis or liver damage or renal impairment.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 257 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Secci, MD, Study Director — Warner Chilcott
Locations (23):
- United States (23):
  - Warner Chilcott Investigational Site, Encino, California
  - Warner Chilcott Investigational Site, Fremont, California
  - Warner Chilcott Investigational Site, Los Angeles, California
  - Warner Chilcott Investigational Site, Sacramento, California
  - Warner Chilcott Investigational Site, Denver, Colorado
  - Warner Chilcott Investigational Site, Miami, Florida
  - Warner Chilcott Investigational Site, Newnan, Georgia
  - Warner Chilcott Investigational Site, Snellville, Georgia
  - Warner Chilcott Investigational Site, Louisville, Kentucky
  - Warner Chilcott Investigational Site, Clinton Township, Michigan
  - Warner Chilcott Investigational Site, Albuquerque, New Mexico
  - Warner Chilcott Investigational Site, Rochester, New York
  - Warner Chilcott Investigational Site, Winston-Salem, North Carolina
  - Warner Chilcott Investigational Site, Cincinnati, Ohio
  - Warner Chilcott Investigational Site, Portland, Oregon
  - Warner Chilcott Investigational Site, Broomall, Pennsylvania
  - Warner Chilcott Investigational Site, Fort Washington, Pennsylvania
  - Warner Chilcott Investigational Site, Austin, Texas
  - Warner Chilcott Investigational Site, College Station, Texas
  - Warner Chilcott Investigational Site, Dallas, Texas
  - Warner Chilcott Investigational Site, Houston, Texas
  - Warner Chilcott Investigational Site, San Antonio, Texas
  - Warner Chilcott Investigational Site, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 4 Mar '08
Groups:
- Doxycycline 0.6 mg/kg/Day: 40 mg doxycycline tablet plus 2 placebo tablets daily
- Doxycycline 1.2 mg/kg/Day: 80 mg doxycycline (1-80 mg tablet) plus 2 placebo tablets daily
- Doxycycline 2.4 mg/kg/Day: 160 mg doxycyline (2-80 mg tablets) plus 1 placebo tablet daily
- Placebo Comparator: 3 placebo tablets daily matching active 40 & 80 mg tablets
Period: Overall Study
Arm/Group | Doxycycline 0.6 mg/kg/Day | Doxycycline 1.2 mg/kg/Day | Doxycycline 2.4 mg/kg/Day | Placebo Comparator
Started | 64 | 65 | 61 | 67
Completed | 52 | 51 | 52 | 54
Not Completed | 12 | 14 | 9 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline 0.6 mg/kg/Day | Doxycycline 1.2 mg/kg/Day | Doxycycline 2.4 mg/kg/Day | Placebo Comparator | Total
Number analyzed (Participants) | 64 | 65 | 61 | 67 | 257
Age Continuous [Mean (Standard Deviation); unit: years] | 19.3 (5.2) | 19.4 (6.6) | 20.7 (7.4) | 20.2 (7.5) | 19.9 (6.7)
Age, Customized [Number; unit: Participants]
  >= 18 years | 32 | 39 | 27 | 35 | 133
  < 18 years | 32 | 26 | 34 | 32 | 124
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 30 | 36 | 35 | 136
  Male | 29 | 35 | 25 | 32 | 121
Region of Enrollment [Number; unit: participants]
  United States | 64 | 65 | 61 | 67 | 257

OUTCOME MEASURES:

1. Primary Outcome: Percentage Patients With Successful Outcome Investigator's Global Assessment (IGA) Score at Week 12, Intent to Treat (ITT) Population
Description: IGA: 0/clear (clear skin no lesions, inflammatory or non-inflammatory), 1/almost clear (rare non-inflammatory lesion w/no more than 1 small inflammatory lesion), 2/mild (some non-inflammatory lesions with no more than a few inflammatory lesions, papules/pustules only, no nodular lesions), 3/moderate (up to many non-inflammatory lesions, some inflammatory lesions, no more than 1 small nodular lesion), 4/severe (many non-inflammatory & inflammatory lesions, no more than a few nodular lesions. Lower score improvement in score. Success=IGA decrease of at least 2 grades from baseline score.
Time Frame: Week 12
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Doxycycline 0.6 mg/kg/Day | Doxycycline 1.2 mg/kg/Day | Doxycycline 2.4 mg/kg/Day | Placebo Comparator
Number analyzed (Participants) | 64 | 65 | 61 | 67
Percentage of Participants | 14.1 [6.6 to 25.0] | 15.4 [7.6 to 26.5] | 29.5 [18.5 to 42.6] | 16.4 [8.5 to 27.5]
Statistical Analysis 1: Comparison: Doxycycline 0.6 mg/kg/Day vs Placebo Comparator; Test type: Superiority or Other; p = 0.779, Cochran-Mantel-Haenszel; Stratified by Investigational Site; Mean Change from Baseline = -0.75, 95% CI 2-sided [-14.8 to 10.3], Standard Deviation 0.85
Statistical Analysis 2: Comparison: Doxycycline 1.2 mg/kg/Day vs Placebo Comparator; Test type: Superiority or Other; p = 0.983, Cochran-Mantel-Haenszel; Stratified by Investigational Site; Mean Change from Baseline = -0.69, 95% CI 2-sided [-13.7 to 11.7], Standard Deviation 0.90
Statistical Analysis 3: Comparison: Doxycycline 2.4 mg/kg/Day vs Placebo Comparator; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel; Stratified by Investigational Site; Mean Change from Baseline = -0.92, 95% CI 2-sided [-1.5 to 27.3], Standard Deviation 0.97

2. Primary Outcome: Absolute Change in Inflammatory Lesion Count From Baseline to Week 12, ITT Population
Description: Change derived as Baseline evaluation minus the Week 12 evaluation. Thus a positive change reflects a reduction in lesion count. Inflammatory Lesion Count includes nodules, papules and pustules.
Time Frame: Baseline to Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Doxycycline 0.6 mg/kg/Day | Doxycycline 1.2 mg/kg/Day | Doxycycline 2.4 mg/kg/Day | Placebo Comparator
Number analyzed (Participants) | 64 | 65 | 61 | 67
Lesions | 8.1 (13.2) | 11.5 (12.1) | 14.0 (19.7) | 7.3 (13.8)
Statistical Analysis 1: Comparison: Doxycycline 0.6 mg/kg/Day vs Placebo Comparator; Test type: Superiority or Other; p = 0.807, Cochran-Mantel-Haenszel; Stratified by Investigational Site
Statistical Analysis 2: Comparison: Doxycycline 1.2 mg/kg/Day vs Placebo Comparator; Test type: Superiority or Other; p = 0.075, Cochran-Mantel-Haenszel; Stratified by Investigational Site
Statistical Analysis 3: Comparison: Doxycycline 2.4 mg/kg/Day vs Placebo Comparator; Test type: Superiority or Other; p = 0.039, Cochran-Mantel-Haenszel; Stratified by Investigational Site

3. Secondary Outcome: Absolute Change From Baseline to Week 12 in NonInflammatory Lesion Count, ITT Population
Description: Noninflammatory Lesion Count includes open and closed comedones.
Time Frame: Baseline to Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Doxycycline 0.6 mg/kg/Day | Doxycycline 1.2 mg/kg/Day | Doxycycline 2.4 mg/kg/Day | Placebo Comparator
Number analyzed (Participants) | 64 | 65 | 61 | 67
Lesions | 8.5 (19.1) | 5.2 (28.1) | 6.5 (16.2) | 1.8 (31.0)
Statistical Analysis 1: Comparison: Doxycycline 0.6 mg/kg/Day vs Placebo Comparator; Test type: Superiority or Other; p = 0.212, Cochran-Mantel-Haenszel; Stratified by Investigational Site
Statistical Analysis 2: Comparison: Doxycycline 1.2 mg/kg/Day vs Placebo Comparator; Test type: Superiority or Other; p = 0.505, Cochran-Mantel-Haenszel; Stratified by Investigational Site
Statistical Analysis 3: Comparison: Doxycycline 2.4 mg/kg/Day vs Placebo Comparator; Test type: Superiority or Other; p = 0.399, Cochran-Mantel-Haenszel; Stratified by Investigational Site

4. Secondary Outcome: Absolute Change From Baseline to Week 12 in Total Lesion Count, ITT Population
Description: Total Lesion Count is the sum of inflammatory and noninflammatory lesions.
Time Frame: Baseline to Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Doxycycline 0.6 mg/kg/Day | Doxycycline 1.2 mg/kg/Day | Doxycycline 2.4 mg/kg/Day | Placebo Comparator
Number analyzed (Participants) | 64 | 65 | 61 | 67
Lesions | 16.6 (25.6) | 16.8 (32.7) | 20.5 (25.0) | 9.1 (38.1)
Statistical Analysis 1: Comparison: Doxycycline 0.6 mg/kg/Day vs Placebo Comparator; Test type: Superiority or Other; p = 0.276, Cochran-Mantel-Haenszel; Stratified by Investigational Site
Statistical Analysis 2: Comparison: Doxycycline 1.2 mg/kg/Day vs Placebo Comparator; Test type: Superiority or Other; p = 0.231, Cochran-Mantel-Haenszel; Stratified by Investigational Site
Statistical Analysis 3: Comparison: Doxycycline 2.4 mg/kg/Day vs Placebo Comparator; Test type: Superiority or Other; p = 0.081, Cochran-Mantel-Haenszel; Stratified by Investigational Site

ADVERSE EVENTS:
Time Frame: 4 Mar 2008 thru 6 Nov 2008
Description: 12 week treatment period for each participant
Arm/Group | Doxycycline 0.6 mg/kg/Day | Doxycycline 1.2 mg/kg/Day | Doxycycline 2.4 mg/kg/Day | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/65 | 0/61 | 1/67
Other Adverse Events (participants affected / at risk) | 22/64 | 20/65 | 29/61 | 25/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline 0.6 mg/kg/Day (N=64) | Doxycycline 1.2 mg/kg/Day (N=65) | Doxycycline 2.4 mg/kg/Day (N=61) | Placebo Comparator (N=67)
Fracture (Left Radius) (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doxycycline 0.6 mg/kg/Day (N=64) | Doxycycline 1.2 mg/kg/Day (N=65) | Doxycycline 2.4 mg/kg/Day (N=61) | Placebo Comparator (N=67)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 2 | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 1 | 2
Fungal Infection (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 6 | 4 | 4 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 8 | 2
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3
Procedural Pain (Nervous system disorders) | 2 | 0 | 1 | 2
Seasonal Allergy (Immune system disorders) | 1 | 0 | 0 | 2
Sunburn (Injury, poisoning and procedural complications) | 0 | 4 | 1 | 1
Toothache (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less